CLINICAL TRIAL: NCT07173647
Title: Pediatric Endurance and Limb Strengthening Program With and Without Electrical Muscle Stimulation Among Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Maryam Iqbal, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0041
Record Dates: First submitted 2025-09-07; First posted 2025-09-15 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy (CP)
Keywords: Pediatric Rehabilitation; Electrical Muscle Stimulation (EMS); Strength Training; Endurance Training; Balance and Gait; Neurorehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Model Description:This study follows a parallel assignment design in which participants are randomly allocated into two groups. Group A will receive the Pediatric Endurance and Limb Strengthening (PEDAL) program combined with Electrical Muscle Stimulation (EMS), while Group B will receive the PEDAL program without EMS. Both groups will be treated and assessed in parallel over the 4-week intervention period
Who Masked: Outcomes Assessor
Masking Description: This study will be conducted as an open-label randomized clinical trial. Due to the nature of the interventions, neither the participants nor the treating physiotherapists can be masked to group allocation. However, to reduce the risk of bias, outcome assessments will be performed by an independent assessor who will not be informed of the group assignments. This approach ensures that data collection remains objective while allowing the interventions to be delivered appropriately.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEDAL Program with Electrical Muscle Stimulation (Experimental): Participants in this group will receive the Pediatric Endurance and Limb Strengthening (PEDAL) program combined with electrical muscle stimulation (EMS) applied to the quadriceps muscles during stationary cycling exercises. Each session will last 60 minutes, three times per week for four weeks, and will include warm-up, strengthening and endurance cycling, and cool-down stretching. EMS parameters will follow established clinical guidelines for strength and endurance training.
  Interventions: Device: PEDAL Program with Electrical Muscle Stimulation
- PEDAL Program without Electrical Muscle Stimulation (Active Comparator): Participants in this group will receive the Pediatric Endurance and Limb Strengthening (PEDAL) program only, without electrical muscle stimulation. The program will also be delivered using stationary cycling for 60 minutes per session, three times per week for four weeks, with warm-up, strengthening and endurance cycling, and cool-down stretching, following the same protocol as the intervention group but without EMS.
  Interventions: Behavioral: PEDAL Program without Electrical Muscle Stimulation

INTERVENTIONS:
Device: PEDAL Program with Electrical Muscle Stimulation — Electrical Muscle Stimulation (EMS) will be applied to the quadriceps muscles of children with cerebral palsy during stationary cycling sessions as part of the Pediatric Endurance and Limb Strengthening (PEDAL) program. EMS will be delivered using clinically approved portable stimulators at parameters appropriate for muscle strengthening and endurance training (frequency 35-50 Hz, pulse width 200-400 μs, duty cycle on/off as tolerated). EMS will be administered simultaneously with cycling to enhance muscle activation and improve motor outcome
  Arms: PEDAL Program with Electrical Muscle Stimulation
Behavioral: PEDAL Program without Electrical Muscle Stimulation — The PEDAL program is a structured exercise intervention designed for children with cerebral palsy. It includes 60-minute sessions of stationary cycling, warm-up, endurance and limb strengthening exercises, and cool-down stretching. Sessions are conducted three times per week for four weeks under therapist supervision. This program is used in both arms of the trial, with or without adjunct Electrical Muscle Stimulation (EMS).
  Arms: PEDAL Program without Electrical Muscle Stimulation

SUMMARY:
This randomized clinical research will assess the impact of a Pediatric Endurance and Limb Strengthening (PEDAL) program, both with and without Electrical Muscle Stimulation (EMS), on balance, gait, and mobility in children diagnosed with cerebral palsy. A total of 26 individuals will be recruited via purposive sampling and randomly allocated to two groups utilizing the sealed envelope method. Group A will undergo the PEDAL program in conjunction with electrical muscle stimulation (EMS) administered to the quadriceps during stationary cycling, whereas Group B will participate in the PEDAL program exclusively, without EMS. Both groups will participate in supervised sessions three times weekly for four weeks, with each session lasting 60 minutes and comprising a warm-up, cycling-based strength and endurance training, and cool-down stretches. EMS parameters will be implemented in accordance with published protocols for strength (30-80 Hz, 150-350 μs) and endurance (8-35 Hz, 150-250 μs) training. Outcome measures, comprising the Berg Balance Scale, Timed Up and Go Test, and Gait Outcomes Assessment List (GOAL™️) questionnaire, will be evaluated at baseline and following four weeks of intervention. The data will be examined utilizing SPSS version 27. This study aims to determine whether incorporating EMS into a structured pediatric strengthening and endurance regimen yields greater improvements in motor function compared to exercise alone.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a predominant cause of childhood impairment, characterized by diminished strength, decreased endurance, inadequate postural control, and restrictions in movement and mobility. Rehabilitation regimens emphasizing endurance and limb strengthening have demonstrated beneficial impacts on motor performance and functional independence in this demographic. Nonetheless, voluntary muscular activation in children with cerebral palsy is frequently constrained, potentially diminishing the efficacy of traditional exercise regimens. Electrical muscle stimulation (EMS) has been implemented as a supplementary method to augment muscle recruitment, reduce stiffness, and enhance neuromuscular control. This trial will examine the Pediatric Endurance and Limb Strengthening (PEDAL) program, both with and without Electrical Muscle Stimulation (EMS), in children diagnosed with cerebral palsy. The PEDAL program employs cycling-based training aimed at enhancing aerobic endurance and lower-limb strength, integrating increasing resistance and functional task elements. In the intervention group, electrical muscle stimulation (EMS) will be administered to the quadriceps muscles during exercise to enhance contractions and potentially increase the training benefits. The study aims to determine if the integration of EMS with endurance and strength training yields superior enhancements in balance, gait, and mobility compared to exercise alone. This project aims to enhance the evidence foundation for pediatric neurorehabilitation, perhaps facilitating the incorporation of EMS-assisted exercise into standard physiotherapy for children with cerebral palsy to optimize motor results and independence.

ELIGIBILITY:
Inclusion Criteria:

* Children from 6 to 10 years old
* Both gender
* Participant with spastic cerebral palsy
* Children who can easily follow verbal directions
* Participant with good and fair one lower limb selective motor control
* Participant who can walk independently
* Participant who lies between 1 to 2 levels of Gross motor function
* People who are willing to participate

Exclusion Criteria:

* Participant who had gone under any neurological surgery, orthopedic surgery or bachlofen pump implant in previous year
* Participant who had serial casting or who use any new orthotics from last 3 months
* Participant with involvement in any exercise, physical therapy, or any sports proceeding within last three months
* Participant who had any serious medical condition like diabetes, seizure, or any cardiac disease
* Participant who are involved in any fitness program that can improve cardio respiratory endurance

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go | Baseline to 4 weeks
  Time (seconds) to stand from a chair, walk 3 meters, turn, return, and sit. Lower times indicate better mobility. Used to determine whether the PEDAL program with or without electrical muscle stimulation produces greater improvement in functional mobility.

SECONDARY OUTCOMES:
Gait Outcomes Assessment List | Baseline to 4 weeks
  Parent-reported questionnaire assessing gait-related function and participation in children with cerebral palsy. Higher scores indicate better function.

OTHER OUTCOMES:
Berg Balance Scale | Baseline to 4 weeks
  Performance-based balance assessment (14 items; 0-56). Higher scores indicate better balance. Used to evaluate change following the interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Naro A, Leo A, Russo M, Casella C, Buda A, Crespantini A, Porcari B, Carioti L, Billeri L, Bramanti A, Bramanti P, Calabro RS. Breakthroughs in the spasticity management: Are non-pharmacological treatments the future? J Clin Neurosci. 2017 May;39:16-27. doi: 10.1016/j.jocn.2017.02.044. Epub 2017 Mar 3. PMID 28262404
- [Result] Ferrari A. From movement to action: a new framework for cerebral palsy. Eur J Phys Rehabil Med. 2019 Dec;55(6):852-861. doi: 10.23736/S1973-9087.19.05845-3. Epub 2019 Sep 24. PMID 31556512
- [Result] Downs (2015) reviewed the Berg Balance Scale, emphasizing its importance in physiotherapy practice.
- [Result] Divita (2024) investigated the effects of high- versus low-frequency whole body vibration on TUG, BBS, and walking performance in chronic stroke patients.
- [Result] Christensen et al. (2019) compared TUG performance in pregnant women with pelvic girdle pain to asymptomatic pregnant and non-pregnant women.
- [Result] Cho et al. (2019) developed a dual-mode feedback-controlled cycling system designed for upper limb rehabilitation in children with cerebral palsy.
- [Result] Bartels EM, Korbo L, Harrison AP. Novel insights into cerebral palsy. J Muscle Res Cell Motil. 2020 Sep;41(2-3):265-267. doi: 10.1007/s10974-020-09577-4. PMID 32065339
- [Result] Armstrong EL, Spencer S, Kentish MJ, Horan SA, Carty CP, Boyd RN. Efficacy of cycling interventions to improve function in children and adolescents with cerebral palsy: a systematic review and meta-analysis. Clin Rehabil. 2019 Jul;33(7):1113-1129. doi: 10.1177/0269215519837582. Epub 2019 Apr 2. PMID 30935240
- [Result] Armstrong EL, Boyd RN, Horan SA, Kentish MJ, Ware RS, Carty CP. Functional electrical stimulation cycling, goal-directed training, and adapted cycling for children with cerebral palsy: a randomized controlled trial. Dev Med Child Neurol. 2020 Dec;62(12):1406-1413. doi: 10.1111/dmcn.14648. Epub 2020 Aug 9. PMID 33146438
- [Result] Anwar, A., Waheed, F., Javaid, A., Zahoor, I. A., Malik, A. N., & Abbas, R. (2023). Normative Values of Berg Balance Scale and Timed Up and Go Test in Elderly Females; A Descriptive Study: Berg Balance Scale in Elderly Females. The Healer Journal of Physiotherapy and Rehabilitation Sciences, 3(6), 617-626.